CLINICAL TRIAL: NCT07317323
Title: Norwegian Spontaneous Coronary Artery Dissection Study (NOR-SCAD Study)
Brief Title: Norwegian Spontaneous Coronary Artery Dissection Study
Acronym: NOR-SCAD
Status: Recruiting | Type: Observational
Sponsor: Oslo University Hospital (Other)
Collaborators: University Hospital, Akershus (Other); Haukeland University Hospital, Bergen, Norway (Unknown); Sorlandet Hospital HF (Other Government); Universitetssykehuset i Nord-Norge HF (Unknown); Ullevaal University Hospital (Other); Helse Stavanger HF (Other Government); St.Olavs Hospital, Trondheim University Hospital, Norway (Unknown)
Responsible Party: Principal Investigator, Mette-Elise Estensen, MD, PhD, Consultant Cardiologist, Oslo University Hospital
Other Study IDs: 853139; ProCardio (Other: Oslo University Hospital)
Record Dates: First submitted 2025-12-05; First posted 2026-01-05 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: SCAD; Myocardial Infarction (MI); Women
Keywords: SCAD NORGE; NOR-SCAD; Spontan Koronar arteriedisseksjon studie; Norwegian Spontaneous Coronary artery dissection study
MeSH Terms: conditions — Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Biobank
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Prospective: SCAD

SUMMARY:
The Norwegian Spontaneous Coronary Artery Dissection Study (NOR-SCAD) is a national, multicenter prospective observational study conducted at major hospitals in Norway. The study investigates risk factors and complications of spontaneous coronary artery dissection (SCAD). Patients aged 18 years or older who are hospitalized with SCAD are recruited during the index hospitalization. Each participant will be followed for 52 weeks with scheduled visits at 8 and 12 weeks and a final phone call at 52 weeks. Evaluations include coronary CT angiography (CTA), cardiac assessments, genetic analyses, blood sampling, structured questionnaires, and a cardiopulmonary exercise test (CPET).

DETAILED DESCRIPTION:
Background: SCAD has emerged as an important cause of myocardial infarction, especially among women under 60 years of age, and is a leading cause of pregnancy-related myocardial infarction. Despite increased awareness over the past two decades, SCAD remains under-recognized, and management varies widely because of limited evidence. Key gaps persist in understanding SCAD etiology, precipitating factors, optimal diagnostic follow-up (including the role of CTA), and the incidence of complications.

Objectives:

Primary objectives: Determine the incidence and types of complications and major adverse cardiac events (MACE) within the first year after SCAD.

Secondary objectives: Evaluate the diagnostic and follow-up utility of coronary CTA.

Methods:

* Multicenter prospective observational cohort study.
* Enrollment period: 2025-2035.
* Study population: Adults (≥18 years) hospitalized with angiographically or imaging-confirmed SCAD at participating hospitals in Norway.
* Follow-up duration: 52 weeks per participant.

Study visits and procedures:

1. Week 1: Acute hospitalization with CT index and blood samples
2. Week 8: CT control
3. Week 12: Comprehensive physical examination with cardiac exams, blood samples, CPET
4. Week 52: Final follow-up phone call to assess clinical events

Endpoints includes major cardiac events (MACE), CTA findings and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Spontaneous coronary artery dissection

Exclusion Criteria:

* Severe kidney failure
* Severe allergic reaction to contrast

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Spontaneous coronary artery dissection
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2035-12-31 (Estimated); Study Completion 2035-12-31 (Estimated)

PRIMARY OUTCOMES:
Major Adverse Cardiac Events | From enrollment to the end of follow-up at 52 weeks
  Recurrent myocardial infarction, extra coronary dissection, stroke/TIA, heart failure,

SECONDARY OUTCOMES:
Assessment of Quality of life | 12 weeks after event
  Quality of life assessed by questionnaire WHO-BREF
CTA | Acute and after 12 weeks
  Computed tomography angiography (CTA) findings

CONTACTS AND LOCATIONS:
Overall Officials: Mette Elise Estensen, MD., PhD, Principal Investigator — ProCardio, Kardiologisk avdeling Rikshospitalet, Oslo Univeristy Hospital
Locations (3):
- Norway (3):
  - Haukeland University Hospital, Bergen
  - Akershus University Hospital, Oslo
  - Rikshospitalet, Oslo University Hospital, Oslo

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- See also: ProCardio Home site — https://www.oslo-universitetssykehus.no/en/avdelinger/hjerte-lunge-og-karklinikken/procardio-center-for-innovation2/
- See also: NOR-SCAD — https://www.oslo-universitetssykehus.no/en/avdelinger/hjerte-lunge-og-karklinikken/procardio-center-for-innovation2/scad-norge/